CLINICAL TRIAL: NCT01225718
Title: Ceftriaxone in Non-neutropenic Fever
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Adam Esbenshade, Assistant Professor of Pediatrics, Vanderbilt University Medical Center
Other Study IDs: VICC PED1061; IRB No. 101020
Record Dates: First submitted 2010-10-15; First posted 2010-10-21 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Histiocytosis; Pediatric Patients With Cancer
MeSH Terms: conditions — Histiocytosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective chart review of all patients cared for at Monroe Carell Jr. Children's Hospital at Vanderbilt including the following:

* patients between 2007-2009 with malignancy, Langerhans cell histiocytosis (LCH) or hemophagocytic lymphohistiocytosis (HLH) and a central venous catheter who were under 23 years of age at time of diagnosis in order to ascertain the associated symptoms, management and outcome of all episodes of non-neutropenic fever.
* to identify a subset of low-risk patients that can be safely managed without use of empiric antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with malignancy, Langerhans cell histiocytosis,or hemophagocytic lymphohistiocytosis from 2007 through 2010
* Under 23 years at time of diagnosis of malignancy, Langerhans cell histiocytosis,or hemophagocytic lymphohistiocytosis
* Treated at Monroe Carell Jr. Children's Hospital at Vanderbilt for aforementioned diagnosis from 2007 through 2012
* While on immunosuppressive therapy with a central venous line in place had at least one documented episode of fever (defined as ≥ 38.0°Celsius orally for over 30 minutes or ≥ 38.3°Celsius orally x1).

Exclusion Criteria:

* Does not meet all inclusion criteria as stated above

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients diagnosed with and treated for malignancy, Langerhans cell histiocytosis ,or Hemophagocytic lymphohistiocytosis between 2007 through 2010 at Monroe Carrell Jr. Children's Hospital at Vanderbilt under the age of 23 at diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 463 (Actual)
Dates: Start 2010-08; Primary Completion 2016-06-25 (Actual); Study Completion 2016-06-25 (Actual)

PRIMARY OUTCOMES:
Incidence of catheter-associated blood stream infections from all episodes of non-neutropenic fever in pediatric oncology, Langerhans cell histiocytosis or Hemophagocytic lymphohistiocytosis patients diagnosed and treated at Vanderbilt | 12 months

SECONDARY OUTCOMES:
Identify risk factors associated with increased risk for catheter-associated blood stream infections in non-neutropenic pediatric oncology and histiocytosis patients with unexplained fever by collecting data for all eligible medical records. | 12 months
  Medical records will be reviewed to identify age of patient at diagnosis and at time of non-neutropenic fever episodes,diagnosis, type of central venous line and number of days in place,all blood cultures obtained during treatment, and dates when last chemotherapy was given, presence of symptoms, lab parameters, presentation to clinic versus emergency room and presence of hemodynamic instability.
Effectiveness of administering empiric cefepime or ceftriaxone in a non-neutropenic oncology or histiocytic patient is estimated, using available microbiologic and antimicrobial susceptibility data from blood cultures | 12 months
  Medical chart is reviewed to collect data if patient received ceftriaxone or other antibiotics, assessment of patient's clinical condition and status of central line, and outcome of blood cultures.

CONTACTS AND LOCATIONS:
Locations (1):
- Monroe Carrell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee, United States